CLINICAL TRIAL: NCT06269614
Title: A Multilevel Approach to Assess the Involvement of Gut Microbiome in Autism and Childhood Stress Regulation
Brief Title: Assessing the Gut Microbiome and Its Association With Pediatric Stress and Cognition
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Gesulla Cavanaugh, Assistant Dean of Research and Assessment, Nova Southeastern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: QOL334829
Record Dates: First submitted 2023-12-11; First posted 2024-02-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder; Adverse Childhood Experiences; Stress Reaction
MeSH Terms: conditions — Autism Spectrum Disorder; Fractures, Stress | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Treatment (Experimental): Pediatric Probiotic Treatment
  Interventions: Dietary Supplement: Probiotic
- No Probiotic Treatment (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Probiotic — Consumption of probiotic with parent- as tolerated for 4 weeks.
  Arms: Probiotic Treatment

SUMMARY:
Using a metabolomics approach in combination with eye-tracking data, this research study proposes to gather evidence from two interrelated body systems (gut and brain) in order to assess how the microbiome is involved in stress modulated symptoms in children with autism and children exposed to repeated stress in comparison to a control group.

DETAILED DESCRIPTION:
The purpose of this study is to find out more about stress in children with autism and those who had negative experiences as children. This will help to find new ways to create therapies against stress on children with autism and those from disadvantaged backgrounds. This study is important because Adverse Childhood Experiences events put children at risk for many health issues. The aims include the examination of the involvement of the microbiome in autistic behaviors and as a modulator and response to stress in the pediatric population.

This study is significant in that many studies point to the gut microbiota as a significant mediator to brain function and behavior, while gut microbiome has been found to play a role in stress mediation. In general, microbiome studies in humans are still minimal and are even more lacking in autism and pediatric research; nonetheless, they have facilitated the evaluation of the potential connection between the microbiome and brain function. For these reasons, this research study is even more relevant in the formation of targeted and feasible strategies to find external and internal factors responsible in the buffering of stress in children from disadvantaged backgrounds, and those with autism.

The children who participate in this study will be assessed at two time points; the second time will be after 4-6 weeks from our first meeting. The parent will make the first appointment with the researcher to allow the child take part of the study. The parent will be given a survey to complete on the child and the parent. The parent will also be provided with a stool collection kit. This kit will be used for them to collect stool sample from the participating child before they come to the first and second appointments with the researcher.

The child will watch a short 2-minute video of a medium stressful scenario followed by a fun video. The child will watch the short video while the researchers evaluate the child's interest through their eye movement with an eye tracker on the computer. The child's heart rate will be measured using a Fingertip Pulse Oximeter.

During the first visit with the researcher, the parent will also receive a coupon and instructions to purchase Garden of Life Children's probiotics at the grocery store if they want their child to incorporate the probiotics in their diet for 4 weeks. They will receive instructions for the child to eat more fruits and vegetables after consulting with the child's pediatrician and/or specialist. The parent can have the researcher's recommended children's probiotics, multivitamins, more fruits and vegetables in the child's diet for 4 weeks before returning to the lab for a second observation. The child will again provide spit and stool after the 4 weeks which will be brought back to the lab during the second appointment.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with Autism
* Children with neurotypical development
* Children in foster care
* Children in homeless shelters
* Children 4-7 years old
* Must be able to watch a short video
* Must be able to consume children's powder probiotics for 4 weeks

Exclusion Criteria:

* Children younger than 4, and older than 7.9 years old.
* Inability to watch a screen
* severe cognitive impairment

Ages: 4 Years to 95 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Enteric Microbiome abundance | 4 weeks
  Increase in gut microbiome abundance (from stool samples) based on values from statistical methods, Analysis of Variance to compare differential abundance analysis.
Enteric Microbiome diversity | 4 weeks
  Increase in gut microbiome diversity in the number of beneficial bacteria in the gut (from stool samples) as measured by α-diversity measures using plot_anova_diversity function in microbiomeSeq package.

SECONDARY OUTCOMES:
Improved response to stressor | 4 weeks
  Improved regulated stress response as assessed by salivary cortisol levels from collected saliva while watching the video stressor and the relaxation video (before the probiotics intervention and after the probiotics intervention). Cortisol levels are measured in ug/dL.
Improved physiological response to stressor | 4 weeks
  Improved physiological response to stressor as measured by pulse rate (bpm) and galvanic skin response (peaks) simultaneously (before and after the probiotics intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Gesulla Cavanaugh, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University College of Nursing, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared based on institutional and IRB approval